CLINICAL TRIAL: NCT02432313
Title: 3-Part Study With 2 6-Period Single Dose Parts (Pt 1, Pt 2 Optional) Followed by a 1-Period Multiple Dose Part (Pt 3) to Evaluate Prototype Modified Release Matrix and Multi Particulate Formulations of Anatabine Citrate to Determine PK
Brief Title: Safety, Tolerability, and Pharmacokinetics of Modified and Immediate Release Anatabine Citrate Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rock Creek Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RCP-PK-002
Record Dates: First submitted 2015-04-28; First posted 2015-05-04 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Pharmacokinetics of Anatabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Modified Release Formulation x (MRx) (Experimental): Various formulations of Modified Release anatabine citrate tablets
  Interventions: Drug: Modified Release Formulation x (MRx)

INTERVENTIONS:
Drug: Modified Release Formulation x (MRx) — Subject receives 1 dose of a MRx and is followed. 7-day washout before dosing with another formulation

SUMMARY:
Parts 1 and 2:

Subjects take 1 dose of various formulations of the study product, and provide samples for pharmacokinetic (PK) analysis after each, with at least 7 days between doses.

Part 3:

Subjects take 2-4 doses of study product or placebo for 6 days, plus 1 additional dose, and provides samples for PK analysis.

DETAILED DESCRIPTION:
Parts 1 and 2:

Subjects will be admitted to the clinic on the day before dosing (Day -1). Subjects will fast overnight and receive the study product in the morning of Day 1 in a non-randomized manner. Subjects will remain onsite until 24 h post-dose and will return to the clinical unit at 36 and 48 h post-dose to provide a sample for PK analysis.

There will be at least a 7-day washout between regimens. Subject will be telephoned 3-5 days after the final dose to ensure his/her ongoing well-being.

Part 3:

Subjects will be admitted to the clinic on the day before dosing (Day -1). Subjects will fast overnight (for Day 1 and Day 7) and receive the study product or placebo on a once, twice, or three times a day regimen in a randomized, double-blind manner. Subjects will remain onsite until 24 h after the final dose (Day 7), leaving the clinic on the morning of Day 8 and returning at 36 and 48 h post last-dose to provide a sample for PK analysis.

Subject will be telephoned 3-5 days after the final dose to ensure his/her ongoing well-being.

ELIGIBILITY:
Inclusion Criteria:

* negative for urinary cotinine
* normal test values for liver function
* provide informed consent

Exclusion Criteria:

* clinically significant abnormal biochemistry, hematology, or urinalysis, as judged by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
PK measures of blood anatabine | 0-2 hrs (every 15 min); 2-6 hrs (every 30 min); 6-12 hr (every 60 min); at 18, 24, 36, and 48 hr

SECONDARY OUTCOMES:
reported adverse events or serious adverse events | immediately post-dose to 5-days post-dose

OTHER OUTCOMES:
measures of pro-inflammatory mediators from stimulated peripheral blood mono-nuclear cells | pre-dose to 12 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Sharan Sidhu, MBChB, MRCS, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Nottingham, United Kingdom